CLINICAL TRIAL: NCT04400851
Title: Sintilimab in the Treatment of Advanced and Refractory Pediatric Malignant Tumors-A Phase I Study
Brief Title: Sintilimab in the Treatment of Advanced and Refractory Pediatric Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yizhuo Zhang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-sen-Sintilimab
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab in advanced childhood cancer patients (Experimental)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Patients were enrolled by the design of phase I study standard. Sintilimab was divided into three dosage levels: 1 mg / kg, 3 mg / kg, and 10 mg / kg. The first level of sintilimab was followed by dose escalation

SUMMARY:
This is a single center, single arm, open-label and phase I clinical study. The standard 3 + 3 group design was performed. Patients were enrolled by the design of phase I study standard. Sintilimab was divided into three dose levels: 1 mg / kg, 3 mg / kg, and 10 mg / kg. Dose escalation was carried out from the first level of sintilimab. The study is to evaluate the safety, including dose limited toxicity (DLT) in the treatment of advanced, recurrent, and refractory childhood cancer.

DETAILED DESCRIPTION:
Malignant tumors are the second leading cause of death in China after accidental casualties, which is consistent with developed countries in Europe and America.

Sintilimab is a human monoclonal antibody against PD-1 receptor which was developed in China. It can block the binding of PD-1 of T-lymphocyte and PD-L1 on the surface of tumor cells, release the immunosuppression of tumor cells on immune cells, making immune cells play the role of anti-tumor cell immunity again and kill tumor cells. In the past, the development of immunocheckpoint drugs mainly focused on adult cancer. Immunocheckpoint inhibition has achieved many successes in the adult population, including metastatic melanoma, non-small cell lung cancer, Hodgkin's lymphoma, bladder cancer and head and neck cancer.

In the past, the development of immunocheckpoint drugs mainly focused on adult cancer. Immunocheckpoint inhibition has achieved many successes in adult population. However, some results of the clinical trials of immunocheckpoint inhibitors in children are also promising especially in Hodgkin's lymphoma.

The investigators aimed to determine the maximum tolerable dose and effectiveness in pediatric malignant tumors, so as to lay the foundation for the future phase II / III clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-18 years old;
2. ECOG PS score: 0-1;
3. Pediatric malignant tumors confirmed by histopathology include Hodgkin's lymphoma, mediastinal large B-cell lymphoma, NK / T-cell lymphoma, nasopharyngeal carcinoma, malignant melanoma, neuroblastoma, hepatoblastoma, sarcoma, brain tumor, etc;
4. Late stage patients who failed to receive standard treatment;
5. There must be at least one measurable lesion defined by RECIST or who standard;
6. Estimated survival time ≥ 6 months;
7. Heart function:

   1. LVEF ≥ 50% by color Doppler echocardiography;
   2. EKG showed no myocardial ischemia;
   3. There was no history of arrhythmia requiring drug intervention before admission;
8. Patients must fully recover from the acute toxicity of all previous anticancer chemotherapy;

   1. Myelosuppression chemotherapy: at least 21 days after the last myelosuppression chemotherapy (42 days if nitrosourea was used in the earlier stage);
   2. Experimental drug or anti-cancer therapy other than chemotherapy: it can not be used within the first 28 days before the planned start of the use of sintilimab, and must be clearly recovered from the clinically significant toxicity of the therapy;
   3. Immunotherapy: at least 42 days after completion of any type of immunotherapy (excluding steroids), including immunocheckpoint inhibitors and tumor vaccines;
   4. X-ray therapy (XRT): at least 14 days after local palliative XRT (small oral area); in case of other substantial bone marrow (BM) irradiation, including pre radioiodinated m-iodobenzidine (131I-MIBG) treatment, at least 42 days must be ended;
   5. Stem cell infusion without total body irradiation (TBI): there is no evidence of active graft-versus-host disease. At least 56 days must elapse after transplantation or stem cell infusion;
9. Patients who have previously received CTLA-4 antibody must meet the following conditions to be admitted to the group

   a) More than 12 weeks after the last administration; b）No history of serious immune related adverse events (CTCAE V4.03 G3 or G4);
10. For patients with known no BM involvement:

    1. Neutrophil absolute count (ANC) ≥ One ×109/L；
    2. Platelet count ≥ one hundred ×109/L；
    3. Hemoglobin ≥ 90 g / L;
11. Liver and kidney function should meet the following standards:

    1. Bilirubin (combined + unconjugated sum) ≤ Two point five * upper limit of normal value (ULN) (corresponding to age), patients who have been confirmed as Gilbert's syndrome can be judged according to the researchers;
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ Two point five ×ULN；
    3. Estimated glomerular filtration rate ≥ 30 ml / min/ one point seven three M2 or serum creatinine (CR) ≤ One point five ×ULN；
12. During the period of participating in the study, be able to follow the outpatient treatment, laboratory monitoring and necessary clinical visits;
13. The parents / guardians of the child or adolescent subjects have the ability to understand, agree and sign the study informed consent form (ICF) and the applicable child consent form before initiating any program related procedures; the subjects have the ability to express their consent (when applicable) with the consent of the parents / guardians.

Exclusion Criteria:

1. Received anti-PD-1 or anti-PD-L1 monoclonal antibody or related pathway targeted drugs;
2. Known to be allergic to PD-1 monoclonal antibody or any of its adjuvants; known to have a history of allergic diseases or severe allergic constitution;
3. Patients with other malignant tumor diseases other than those treated by the Institute, except for patients who has been cured and with no recurrence within 3 years before the study was selected, completely removed basal cell and squamous cell skin cancer, completely removed any type of carcinoma in situ;
4. Active central nervous system metastasis (whether or not treated), including symptomatic brain metastasis or meningeal metastasis or spinal cord compression, etc.; except: asymptomatic brain metastasis (no progress within at least 4 weeks after radiotherapy and / or no neurological symptoms or signs after surgical resection, no need for dexamethasone or mannitol treatment).
5. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
6. The toxicity of previous treatment is still more than grade 1 (CTCAE V4.03 Standard), except hair loss and neurotoxicity;
7. Having a history of mental disorders;
8. Those who have a history of drug use or drug abuse upon inquiry;
9. History of idiopathic pulmonary fibrosis or pneumonia;
10. The complications that need to be treated with immunosuppressive drugs, or the complications that need to be treated with systemic or local corticosteroids according to the dose with immunosuppressive effect (prednisone > 10 mg / day or equivalent dose of similar drugs).
11. Have a history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc., except for: type I diabetes, hypothyroidism that can be controlled only through hormone replacement therapy, skin diseases that do not need systemic treatment (such as vitiligo, psoriasis), controlled celiac disease, or Disease that does not recur without external stimulus;
12. Patients with active TB infection before or now;
13. Active infection requiring systemic treatment;
14. Uncontrolled hypertension (systolic ≥ 140 mmHg and / or diastolic ≥ 90 MmHg) or pulmonary hypertension or unstable angina pectoris; myocardial infarction or bypass or stent operation within 6 months before administration; history of chronic heart failure meeting NYHA level 3-4; valvular disease of clinical significance; serious arrhythmia requiring treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia), including QTc interval male ≥ 450ms , female ≥ 470ms (calculated by friderica formula), cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration, etc;
15. Serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc;
16. Anti HIV, TP AB and HCV AB were positive, HBV AG was positive and HBV DNA copy number was higher than the upper limit of normal value of detection unit;
17. Thyroid function was abnormal (FT3, FT4, T3, T4);
18. Major surgery is expected within 28 days before administration or during treatment;
19. Live vaccine or attenuated vaccine is expected to be given 4 weeks before administration, during treatment or within 5 months after the last administration;
20. Participate in another clinical trial and receive the trial drug treatment within 30 days before administration;
21. According to the judgment of the investigator, patients who are not suitable for the trial due to other reasons.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) | From date of enrollment until the end of 1 cycle of treatment, assessed up to 3 weeks
  Determine the appropriate dose of maximum tolerable dose (MTD) of sintilimab for further clinical study in this patient population

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  Hematology and non-hematology toxicity (NCI CTCAE v5.0 )
Objective presponse rate (ORR) | From the date of the treatment to the first evaluation (After 2 cycles of treatment assessed up to 6 weeks)
  complete release and partial release

CONTACTS AND LOCATIONS:
Locations (1):
- Yizhuo Zhang, Guangzhou, China

REFERENCES:
- [Derived] Que Y, Wang J, Sun F, Wang S, Zhu J, Huang J, Zhao Z, Zhang L, Liu J, Xu J, Zhen Z, Sun X, Lu S, Zhang Y. Safety and clinical efficacy of sintilimab (anti-PD-1) in pediatric patients with advanced or recurrent malignancies in a phase I study. Signal Transduct Target Ther. 2023 Oct 13;8(1):392. doi: 10.1038/s41392-023-01636-9. PMID 37828033